CLINICAL TRIAL: NCT00783614
Title: The Effect of Aspirin and Antiretroviral Therapy on Cardiovascular Risk in HIV Infected Patients: A Pilot Study
Brief Title: Aspirin and Antiretroviral Therapy in HIV Infected Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: PCC-002
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection
Keywords: HIV; Cardiovascular Disease; Endothelial Dysfunction
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases | interventions — Aspirin; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Start antiretroviral therapy (ART) immediately and initiate aspirin 325mg po daily
  Interventions: Drug: Aspirin 325mg; Drug: Antiretroviral therapy (ART)
- 2 (Placebo Comparator): Start antiretroviral therapy (ART) immediately and initiate placebo pill daily
  Interventions: Drug: Antiretroviral therapy (ART)
- 3 (Active Comparator): Defer antiretroviral therapy (ART) for 1 month and immediately initiate aspirin 325mg po daily
  Interventions: Drug: Aspirin 325mg; Drug: Antiretroviral therapy (ART)
- 4 (Placebo Comparator): Defer antiretroviral therapy (ART) for 1 month and immediately initiate placebo pill daily
  Interventions: Drug: Antiretroviral therapy (ART)

INTERVENTIONS:
Drug: Aspirin 325mg — Patients randomized to Aspirin 325mg po daily versus placebo pill daily
  Arms: 1; 3
Drug: Antiretroviral therapy (ART) — Patients randomized to start ART immediately or defer use for 1 month

SUMMARY:
The purpose of this study is to examine the effects of HIV treatment (antiretroviral therapy) and aspirin use on risk for cardiovascular disease among HIV infected persons.

DETAILED DESCRIPTION:
Cardiovascular disease is now a major health concern among persons with HIV infection. Our general hypothesis is that HIV-mediated inflammation and injury to vascular surfaces up-regulates thrombotic pathways and leads to damage of blood vessels that is promotes development of cardiovascular disease. HIV drug treatment (antiretroviral therapy; ART) may reduce inflammation and vessel injury via suppression of HIV replication, but also includes side effects or toxicity that may increase risk for cardiovascular disease in and of itself. In this context, additional anti-inflammatory and anti-thrombotic medications are needed. Acetylsalicylic acid (aspirin) is an excellent candidate and is commonly used for secondary prevention of cardiovascular events in the general population, but few studies have examined it's use in persons with HIV infection. The goal of this study is to generate pilot data regarding changes in measures of cardiovascular risk, as determined by reductions in inflammatory and thrombotic blood markers and a decrease in blood vessel injury (blood markers) and dysfunction (assessment of arterial elasticity), that occur after starting ART and aspirin among persons with HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected (by positive HIV Ab or detectable HIV RNA level)
2. No ART for at least previous 3 months
3. Ready to start or re-start ART (regimen pre-chosen by patient and provider)

Exclusion Criteria:

1. Age < 18 years, or >60 years
2. Pregnancy
3. Current aspirin use
4. Presence of known atherosclerotic CVD determined by:

   1. Previous myocardial infarction
   2. Significant coronary atherosclerosis by angiography
   3. Coronary revascularization procedure (coronary stent or surgical bypass)
   4. Previous cerebral vascular accident (stroke)
   5. Ischemic cardiomyopathy
   6. Carotid stenosis (>25% narrowing by carotid ultrasound)
   7. Aortic aneurysm
   8. Symptomatic peripheral vascular disease (claudication)
   9. Surgical revascularization procedure of peripheral vessels
5. Hospitalization (within prior 2 weeks of study entry)
6. Concurrent self-limited bacterial infections (does not include chronic viral infections)
7. Clinical or pathologic diagnosis of systemic vasculitis
8. Active drug or alcohol use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason V Baker, MD, MS, Principal Investigator — University of Minnesota; HCMC
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kunisaki KM, Quick H, Baker JV. HIV antiretroviral therapy reduces circulating surfactant protein-D levels. HIV Med. 2011 Oct;12(9):580-1. doi: 10.1111/j.1468-1293.2011.00920.x. No abstract available. PMID 21951596

RESULTS

PARTICIPANT FLOW:
Groups:
- ART and Aspirin: Start ART immediately and initiate aspirin 325mg po daily
- ART and Placebo: Start ART immediately and initiate placebo pill daily
- Defer and Aspirin: Defer ART for 1 month and immediately initiate aspirin 325mg po daily
- Defer and Placebo: Defer ART for 1 month and immediately initiate placebo pill daily
Period: Overall Study
Arm/Group | ART and Aspirin | ART and Placebo | Defer and Aspirin | Defer and Placebo
Started | 6 | 6 | 5 | 5
Completed | 6 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ART and Aspirin | ART and Placebo | Defer and Aspirin | Defer and Placebo | Total
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 5 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (9.0) | 38.4 (10.6) | 36.0 (9.3) | 37.5 (11.1) | 37.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2 | 4
  Male | 6 | 4 | 5 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 5 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side Effects (Self-report) Number of Participants With Adverse Events
Description: At each visit participants were asked if they were experience side effects to study medications. They were also asked if any new events or symptoms occurred since the last visit, even if they did not suspect it was related to the study medication
Time Frame: 6 months
Population: The number of participants with adverse events or reporting side effects
Measure: Number; unit: participants
Arm/Group | ART and Aspirin | ART and Placebo | Defer and Aspirin | Defer and Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 5
participants | 1 | 0 | 1 | 0

2. Primary Outcome: Blood Markers of Inflammation, Endothelial Injury, and Thrombosis
Time Frame: changes from baseline to 6 months
Population: Data measurements not obtained, as study terminated early due to poor enrollment
Arm/Group | ART and Aspirin | ART and Placebo | Defer and Aspirin | Defer and Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | ART and Aspirin | ART and Placebo | Defer and Aspirin | Defer and Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed. Study recruitment difficulty due to inclusion of ART deferral component.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes